CLINICAL TRIAL: NCT00002098
Title: Phase I/II Study of the Tolerance and Efficacy of Combined Use of Didanosine (2',3'-Dideoxyinosine; ddI) and Lentinan in HIV-Positive Patients
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AJI Pharma USA (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Model: Parallel | Purpose: Treatment
Other Study IDs: 126A; 91-10-15
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1995-03

CONDITIONS: HIV Infections
Keywords: Didanosine; Drug Therapy, Combination; Acquired Immunodeficiency Syndrome; AIDS-Related Complex; Lentinan
MeSH Terms: conditions — HIV Infections; Acquired Immunodeficiency Syndrome; AIDS-Related Complex | interventions — Lentinan; Didanosine

INTERVENTIONS:
Drug: Lentinan
Drug: Didanosine

SUMMARY:
To determine the tolerance and side effects of a combination of lentinan and didanosine (ddI) compared with ddI alone. To determine whether the combination of lentinan and ddI produces a significant immunorestorative effect within the study observation period (6-12 months) as measured by an increase in one or more of the following: neutrophil count and activity, T-cell subsets, and a decrease in p24 antigen.

DETAILED DESCRIPTION:
Patients are randomized to receive either lentinan (40 patients) or placebo (10 patients) in combination with ddI for at least 26 weeks; those tolerating their dose may be offered continuation of therapy for an additional 26 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV seropositivity.
* Absolute CD4 count of 200 - 500 cells/mm3.
* No active opportunistic infection or Kaposi's sarcoma.

Prior Medication:

Allowed:

* Prior ddI for no longer than 3 months.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Lymphoid malignancy.
* Pancreatitis.
* Peripheral neuropathy.
* Critical illness.

Concurrent Medication:

Excluded:

* Antiretroviral agents other than ddI.
* Steroids.
* Cytotoxic agents.
* Immunosuppressive agents.
* Immunomodulators.
* 1-Thyroxine.

Concurrent Treatment:

Excluded:

* Radiotherapy.

Prior Medication:

Excluded within 1 month prior to study entry:

* Antiretroviral agents other than ddI (patients may have received prior ddI for no longer than 3 months total).
* Steroids.
* Cytotoxic agents.
* Immunosuppressive agents.
* Immunomodulators.

Prior Treatment:

Excluded:

* Radiotherapy within 1 month prior to study entry. Active drug abuse.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50

CONTACTS AND LOCATIONS:
Overall Officials: Lang W, Study Chair; Goodgame J, Study Chair
Locations (2):
- United States (2):
  - ViRx Inc, San Francisco, California
  - Goodgame Med Group, Maitland, Florida

REFERENCES:
- [Background] Gordon M, Guralnik M, Kaneko Y, Mimura T, Goodgame J, DeMarzo C, Pierce D, Baker M, Lang W. A phase II controlled study of a combination of the immune modulator, lentinan, with didanosine (ddI) in HIV patients with CD4 cells of 200-500/mm3. J Med. 1995;26(5-6):193-207. PMID 8721897
- [Background] Kaneko Y, Mimura T, Guralnik M, Baker M, Goodgame J, DeMarzo C, Pierce D, Lang W, Gordon M. Phase II study of combination of lentinan with ddI in HIV-positive patients. Int Conf AIDS. 1994 Aug 7-12;10(1):212 (abstract no PB0276)